CLINICAL TRIAL: NCT05837247
Title: Effects of Telemonitoring-supported Game-based Home Exercises on Kinesiophobia, Pain and Quality of Life in Juvenile Idiopathic Arthritis
Brief Title: Effects of Telemonitoring-supported Game-based Home Exercises in Juvenile Idiopathic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gokce Leblebici, Asssistant professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulUC_ccrpts
Record Dates: First submitted 2023-03-29; First posted 2023-05-01 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Exercise Therapy; Juvenile Idiopathic Arthritis
Keywords: telemonitoring; physiotherapy; juvenile idiopathic arthritis; game-based exercises; telerehabilitation; remote methods
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game-based telerehabilitation exercises (Experimental): The telemonitoring-supported program will be conducted with a smartphone application synchronously. The participants will be monitored by the investigators using an online communication application during exercise sessions.The sessions will be conducted to patients' individual calender via a smartphone application and a reminder from this smartphone application will send notifications to the patients.
  Interventions: Other: Game-based telerehabilitation exercises
- Control group (Active Comparator): The control group will be evaluated and followed with home exercise program.
  Interventions: Other: Home exercises

INTERVENTIONS:
Other: Game-based telerehabilitation exercises — online Game-based home exercises are physiotherapy programs that include exercises transformed into game activities to increase the child's participation in the rehabilitation process. The exercises were planned such as; the dwarf camel game as squat exercises; the flamingo balance game as single leg balance exercises and weight-bearing activities etc. The exercise program will be conducted for 6 weeks and 3 sessions in a week.
  Arms: Game-based telerehabilitation exercises
Other: Home exercises — The physiotherapist will evaluate the control group patients and monitor them using only a home exercise program.
  Arms: Control group

SUMMARY:
In order to cope with pain, improve quality of life and prevent kinesiophobia in children with juvenile idiopathic arthritis, most of the physiotherapy approaches used so far are standard.

However, nowadays, it has been observed that participation in treatment has increased with game-based exercises instead of standard physiotherapy. In addition, remote monitoring applications made it possible to perform physiotherapy programs, which are an integral part of the treatment in children with JIA, who is difficult to reach the clinic due to reasons such school schedule and living area, through remote monitoring. This project aimed to investigate the effects of telemonitoring-supported game-based home exercise programs on pain, kinesiophobia and quality of life.

The original aspect of our project is to include telemonitoring-supported game-based home exercise programs as an alternative physiotherapy program in children with JIA. Its contribution to clinical practice is to change the perspective of physiotherapists and children on standard physiotherapy practices, to increase their motivation, and to ensure children's participation in treatment.

DETAILED DESCRIPTION:
Juvenile rheumatic diseases are chronic diseases with a prognosis ranging from complete recovery to long-term disability. Juvenile idiopathic arthritis (JIA) is the most common rheumatologic disease in children. Pain is one of the main clinical symptoms in JIA. Due to pain, these children with rheumatic diseases avoid moving. The fear of moving because of this pain is defined as kinesiophobia. Kinesiophobia (fear of movement); It is defined as an excessive and unreasonable fear of physical action to avoid harm or re-injury. Its prevalence in chronic pain varies between 50-70%. Regular physical activity and fitness exercises can prevent kinesiophobia; Treatment includes therapeutic exercises and cognitive behavioral therapy.

In order to cope with pain, improve quality of life and prevent kinesiophobia in children with juvenile idiopathic arthritis, most of the physiotherapy approaches used so far are standard.

However, nowadays, it has been observed that participation in treatment has increased with game-based exercises instead of standard physiotherapy. In addition, remote monitoring applications made it possible to perform physiotherapy programs, which are an integral part of the treatment in children with JIA, who is difficult to reach the clinic due to reasons such school schedule and living area, through remote monitoring. This project aimed to investigate the effects of telemonitoring-supported game-based home exercise programs on pain, kinesiophobia and quality of life.

In this study, the participants will be evaluated and training game-based exercises at the baseline examination. Then, the participants will be followed the online synchronous communication application-based telemonitoring method After the game-based home exercises intervention, the participants will be re-evaluated again and the results will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Whose are diagnosed with JIA at least 1 year ago
2. Whose are aged 6-16 years
3. Whose are having pain in lower extremity joints for more than the last 6 months
4. Whose have stable medical treatment
5. Whose are at a level to understand the games and perform the activities mentally

Exclusion Criteria:

1. Patients with neurological problems in addition to rheumatic diagnosis
2. Individuals who are contraindicated to exercise

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
The Wong-Baker Faces Pain Rating Scale | immediately After intervention
  A self-report tool called The Wong-Baker Faces Pain Rating Scale is used to assess how much pain kids are experiencing. It is widely acknowledged that measuring children's pain is challenging for medical professionals.
  This is because children express pain differently than adults due to differences in their language, communication, and developmental stages.
  The Wong-Baker Pain Scale has 6 faces. The first face represents a pain score of 0 and indicates "not hurt". The second face is a 2 represents the pain score and means "it hurts a little". The third face represents a pain score of 4 and "it hurts a little more" shows. The fourth face represents a pain score of 6 and indicates "it hurts more". The fifth face represents a pain score of 8.
  and shows that "it hurts a lot"; the sixth face represents a pain score of 10 and indicates "worst pain". The unit of this outcome is a score.
Pediatric Quality of Life Inventory (PedsQL) 3.0 Arthritis Module | immediately After intervention
  Patients with JIA have the Pediatric Quality of Life Inventory (PedsQL) 3.0 arthritis module. This criterion has been translated into Turkish and its validity has been demonstrated. 44 Evaluations are made about pain and suffering (four questions), daily activities (five questions), treatment (seven questions), anxiety (three questions), communication (three questions), and parent and child modules are evaluated separately. The unit of this outcome is a score. Every item is 5-point Likert scale type. Scores are transformed on a scale from 0 to 100. Items are reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Higher scores mean better quality of life and fewer problems or symptoms
The Tampa Scale for Kinesiophobia | immediately After intervention
  It is a 17-item scale developed to measure the fear of movement/re-injury. The scale includes parameters of injury/re-injury and fear-avoidance in work-related activities. A 4-point Likert scoring (1 = I strongly disagree, 4 = I totally agree) is used in the scale. After reversing items 4, 8, 12 and 16, a total score is calculated. The person gets a total score between 17-68. A high score on the scale indicates a high level of kinesiophobia. It is recommended to use the total score in studies. In our study, the fear of avoiding movement will be evaluated with TSK. The unit of this outcome is a score.
Hip flexion-extension range of motion | immediately After intervention
  The pre-study and post-study hip flexion/extension passive ranges of motion (ROM) were measured by goniometric measurement.
Hip internal-external rotation range of motion | immediately After intervention
  The pre-study and post-study hip internal-external rotation passive ranges of motion (ROM) were measured by goniometric measurement.
Hip abduction/adduction range of motion | immediately After intervention
  The pre-study and post-study hip abduction/adduction passive ranges of motion (ROM) were measured by goniometric measurement.
Knee flexion and extension range of motion | immediately After intervention
  The pre-study and post-study knee flexion and extension passive ranges of motion (ROM) were measured by goniometric measurement.
Ankle dorsi-plantar flexion range of motion | immediately After intervention
  The pre-study and post-study ankle dorsi-plantar flexion passive ranges of motion (ROM) were measured by goniometric measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Gökçe Leblebici, Phd, Pt, Study Chair — Istanbul Medeniyet University
Locations (1):
- İstanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crayne CB, Beukelman T. Juvenile Idiopathic Arthritis: Oligoarthritis and Polyarthritis. Pediatr Clin North Am. 2018 Aug;65(4):657-674. doi: 10.1016/j.pcl.2018.03.005. PMID 30031492
- [Background] Arman N, Tarakci E, Tarakci D, Kasapcopur O. Effects of Video Games-Based Task-Oriented Activity Training (Xbox 360 Kinect) on Activity Performance and Participation in Patients With Juvenile Idiopathic Arthritis: A Randomized Clinical Trial. Am J Phys Med Rehabil. 2019 Mar;98(3):174-181. doi: 10.1097/PHM.0000000000001001. PMID 30020092
- [Background] Minden K, Niewerth M. [Juvenile idiopathic arthritis--clinical subgroups and classification]. Z Rheumatol. 2008 Mar;67(2):100, 102-6, 108-10. doi: 10.1007/s00393-007-0246-5. German. PMID 18299857
- [Background] Weermeijer JD, Meulders A. Clinimetrics: Tampa Scale for Kinesiophobia. J Physiother. 2018 Apr;64(2):126. doi: 10.1016/j.jphys.2018.01.001. Epub 2018 Mar 19. No abstract available. PMID 29567379
- [Background] Zaripova LN, Midgley A, Christmas SE, Beresford MW, Baildam EM, Oldershaw RA. Juvenile idiopathic arthritis: from aetiopathogenesis to therapeutic approaches. Pediatr Rheumatol Online J. 2021 Aug 23;19(1):135. doi: 10.1186/s12969-021-00629-8. PMID 34425842
- [Background] Grassini S. Virtual Reality Assisted Non-Pharmacological Treatments in Chronic Pain Management: A Systematic Review and Quantitative Meta-Analysis. Int J Environ Res Public Health. 2022 Mar 29;19(7):4071. doi: 10.3390/ijerph19074071. PMID 35409751
- [Background] Hadjiat Y, Marchand S. Virtual Reality and the Mediation of Acute and Chronic Pain in Adult and Pediatric Populations: Research Developments. Front Pain Res (Lausanne). 2022 May 6;3:840921. doi: 10.3389/fpain.2022.840921. eCollection 2022. PMID 35599969
- [Derived] Leblebici G, Kisa EP, Tarakci E, Gunhan I, Yenici EN, Kasapcopur O. Gamified Telerehabilitation in Oligoarticular Juvenile Idiopathic Arthritis: A Randomized Controlled, Single-Blind Trial. Int J Rheum Dis. 2025 Jul;28(7):e70342. doi: 10.1111/1756-185X.70342. PMID 40631545